CLINICAL TRIAL: NCT02585401
Title: Evaluation of Physician Knowledge of Key Safety Information for Eylea in Canada: An Observational Postauthorization Safety Study
Brief Title: Evaluation of Physician Knowledge of Safety and Safe Use Information for Aflibercept in Canada
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 18498
Record Dates: First submitted 2015-10-22; First posted 2015-10-23 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Age-related Macular Degeneration (AMD); Central Retinal Vein Occlusion (CRVO); Diabetic Macular Edema (DME)
MeSH Terms: conditions — Macular Degeneration; Retinal Vein Occlusion | interventions — aflibercept

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Eylea product and application information / Cohort 1: Physicians prescribing aflibercept in Canada will be selected to reflect the distribution of retinal specialists and ophthalmologists who prescribe aflibercept.
  Interventions: Drug: Eylea (Aflibercept, VEGF Trap-Eye, BAY86-5321)

INTERVENTIONS:
Drug: Eylea (Aflibercept, VEGF Trap-Eye, BAY86-5321) — The physician questionnaire will contain primarily closed-ended questions (e.g., multiple choice, true/false), with few free-text response fields, eliciting responses measuring physician knowledge and understanding of the key information in the Eylea vial preparation instruction card, the intravitreal injection procedure video, and the product monograph.

SUMMARY:
The primary objective of this study is to measure physician knowledge and understanding of the key safety information contained in the Eylea vial preparation instruction card, the intravitreal injection procedure video, and the product monograph.

DETAILED DESCRIPTION:
The source of information for the study will be self-reported data collected from physicians using standard questionnaires with closed-ended response choices. Questionnaires for physicians will be developed and tested using best practices for instrument development. The questions will be tailored to the study aims and the information provided in the the vial preparation instruction card, the intravitreal injection procedure video, and the Eylea product monograph.

Other questions will obtain information needed to assess potential differences across subgroups and identify any biases (e.g., demographics, experience with Eylea).

The questionnaire will be tested through cognitive interviews with physicians. Questionnaires will be tested in local languages, to assure that the introductory material, consent forms, and questionnaire items (question stems and response choices) are culturally appropriate and easily and correctly understood by individuals similar to those who will participate

ELIGIBILITY:
Inclusion Criteria:

This study will be conducted with retinal specialists and ophthalmologists in Canada who have prescribed and/or administered aflibercept to at least 1 patient in the past 6 months.

Exclusion Criteria:

* None applied

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Physicians prescribing aflibercept in Canada will be selected to reflect the distribution of retinal specialists and ophthalmologists who prescribe aflibercept.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2016-02-18 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-05-19 (Actual)

PRIMARY OUTCOMES:
Knowledge and understanding of key information contained in the aflibercept educational materials: the Eylea vial preparation instruction card, the intravitreal injection procedure video, and the product monograph | Up to 8 weeks after the start of data collection
  The source of information for the study will be self-reported data collected from physicians using standard questionnaires with closed-ended response choices.

SECONDARY OUTCOMES:
Investigation whether physicians have received the educational materials | up to 6 month
  Descriptive results assessing Number and percentage (%) of physicians

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Canada